CLINICAL TRIAL: NCT06615024
Title: Newborn Screening of Coexistence Between Sickle Cell Anaemia and G6PD Deficiency in NEW VALLEY GOVERNORATE
Brief Title: Screening of Coexistence Between Sickle Cell Anaemia and G6PD Deficiency
Status: Not yet recruiting | Type: Observational
Sponsor: Fatma Hussein Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Fatma Hussein Mahmoud, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Coexistence of SCD and G6PD
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Sickle Cell Disease and G6PD Deficiency
MeSH Terms: conditions — Anemia, Sickle Cell; Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — EDTA samples and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Newborns who are delivered in NEW VALLEY GOVERNORATE: Screening of coexistence between sickle cell anaemia and G6PD deficiency
  Interventions: Diagnostic Test: G6pd enzyme sickling test; Diagnostic Test: G6PD enzyme and sickling test; Diagnostic Test: G6PD enzyme and HPLC

INTERVENTIONS:
Diagnostic Test: G6pd enzyme sickling test — Measuring the enzyme level of G6PD and presence of Hbs
Diagnostic Test: G6PD enzyme and sickling test — Measuring enzyme level of G6PD and level of HbS
Diagnostic Test: G6PD enzyme and HPLC — Measuring G6PD enzyme level in neonates and measuring level of HbS

SUMMARY:
G6PD deficiency may have a subtle effect on the severity of hemolysis and also worsen the degree of anaemia in SCD when the two disorders coexist. Therefore, selective decision should be taken in patients in whom the two conditions coexist in the choice of drug and in the treatment of infections.The prevalence of the G-6-PD deficiency is high in SCD patients, but does not differ from that observed among non-SCD subjects .However, the G-6-PD deficiency appears to worsen the clinical features of SCD, there were more hospitalizations, major vaso-occlusive crises among G-6-PD deficient sickle cell patients.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is not frequent in Egypt except in the Oases where the carrier rate varies from 9 to 22%. It is a hereditary blood disorder characterized by the production of abnormal hemoglobin molecules that cause red blood cells to take on a crescent or sickle shape. This haemoglobin called haemoglobin S, which causes red blood cells to become stiff and sticky, leading to various health complications as recurrent pain, fatigue, anaemia, and increased infection susceptibility.prevalence of G6PD deficiency is 4.3% with a male:female ratio of 3.2:1. Enzyme activity was significantly higher in males than females. It is located on X chromosome which leads to a lower level of reduced glutathione, an antioxidant, in red blood cells (RBCs). Most of the time, those who are affected have no symptoms. However, they should avoid specific triggers that may promote oxidative stress such as fava beans, that may fragilize RBCs and cause hemolysis. G6PD deficiency may have a subtle effect on the severity of hemolysis and also worsen the degree of anaemia in SCD when the two disorders coexist. Therefore, selective decision should be taken in patients in whom the two conditions coexist in the choice of drug and in the treatment of infections. The prevalence of the G-6-PD deficiency is high in SCD patients, but does not differ from that observed among non-SCD subjects .However, the G-6-PD deficiency appears to worsen the clinical features of SCD, there were more hospitalizations, major vaso-occlusive crises among G-6-PD deficient sickle cell patients.

ELIGIBILITY:
Inclusion Criteria:

- All new born with good general health

Exclusion Criteria:

* 1-new born with high reticulocytic count 2-new born with bad general health

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted on all newborn delivered in pediatric department in NEW VALLEY UNIVERSITY from jan2025 to Jan 2026
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
prevelance of coexistence between sickle cell anaemia and G6PD deficiency in NEW VALLEY GOVERNORATE | One year
  Evaluate the prevalence of coexistence between sickle cell anaemia and G6PD deficiency in NEW VALLEY GOVERNORATE to create data base for endemic hereditary disease

SECONDARY OUTCOMES:
Early diagnosis to decrease incidanc of complications | One year
  Early diagnosis of coexistence between sickle cell anaemia and G6PD deficiency to tell specific treatment and maintain haemoglobin level high to prevent more complications